CLINICAL TRIAL: NCT03525015
Title: Impact of a Printed Decision Aid on Cataract Surgery Choice: A Multi-center Randomized Controlled Trial
Brief Title: Impact of a Printed Decision Aid on Cataract Surgery Choice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Clinical investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017KYPJ066
Record Dates: First submitted 2018-04-12; First posted 2018-05-15 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Age Related Cataracts
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A decision aid booklet (Experimental): A decision aid booklet about cataract surgery choice
  Interventions: Other: A decision aid booklet about cataract surgery choice
- An usual booklet (Active Comparator): An usual booklet about cataract and cataract surgery
  Interventions: Other: An usual booklet about cataract and cataract surgery

INTERVENTIONS:
Other: A decision aid booklet about cataract surgery choice — Potential participants receive a decision aid booklet with information about cataract surgery choice, and outcome data will be gathered using standardized questions in a structured interview after 2 weeks and 1 year.
  Arms: A decision aid booklet
Other: An usual booklet about cataract and cataract surgery — Potential participants receive an usual booklet with information about cataract and cataract surgery, and outcome data will be gathered using standardized questions in a structured interview after 2 weeks and 1 year.
  Arms: An usual booklet

SUMMARY:
The purpose of the study is to explore whether a decision aid booklet is more effective than the usual booklet for patients to make an informed choice on cataract surgery.

DETAILED DESCRIPTION:
Shared decision making is increasingly recommended to facilitate quality care, but there is a lack of cataract surgery decision aid in clinical practice. The aim of this study is to evaluate the effectiveness of a cataract surgery decision aid for cataract patients with different levels of health literacy.

We will conduct a randomized controlled trial for cataract patients aged 50-80 years. We will randomly assign participants to either the intervention using a decision aid booklet or the one using a usual cataract booklet. The primary outcome is informed choice (defined as adequate knowledge and consistency between attitudes and intentions) 2 weeks after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis of age-related cataract;
2. The best corrected visual acuity (BCVA) is above 20/60;
3. Cataract opacity meets any of the following criterion based on lens opacity classification system (LOCS) III: nuclear color and nuclear opalescence is greater than or equal to grade 2 (NO2/NC2); cortical opacity is greater than or equal to grade 2 (C2); posterior subcapsular opacity is greater than or equal to grade 2 (P2);
4. Willing to know about cataract and cataract surgery;
5. Being able to afford cataract surgery;
6. Willing to participate in the study and provide the informed content.

Exclusion Criteria:

1. Having received cataract surgery;
2. Having hearing disorders;
3. Having mental disorders;
4. Having ocular disorders other than cataract;
5. Having surgery contraindication;
6. Unwilling to participate in this study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Informed choice about cataract surgery | 2 weeks
  Informed choice is measured as the proportion of participants who make an informed choice about whether to receive cataract surgery as soon as possible or not. For the individual, making an informed choice is defined as (i) having adequate knowledge and (ii) expressing intentions that are consistent with （iii）one's attitudes. Knowledge will be measured by assessing participants' understanding of the numerical and conceptual information in the booklets, using items modified from previous screening decision aid trials (Hersch 2015). Attitudes towards cataract surgery will be assessed using a theory-based generic screening attitudes scale (Dormandy 2006). A single item will measure intentions about having cataract surgery as soon as possible (or not), using a set of 5 response options (Gwyn 2003; Watson 2006).

SECONDARY OUTCOMES:
Perceived importance of cataract surgery benefit/harms | 2 weeks
  Purpose-developed items will be used to ask participants about their personal perceptions of the importance of specific outcomes in their decision-making about cataract surgery. Participants will be asked how important it is to (i) have significant increase in vision-related quality of life, and (ii) have no significant increase in vision-related quality of life after receiving cataract surgery as soon as possible. The four response options range from very important to not at all important (Hersch 2014).
Perceived personal chances of surgical benefit/harms | 2 weeks
  Participants will be asked about their perceived personal likelihood of experiencing specific outcomes if they have cataract surgery as soon as possible, compared with an average patient who had undergone cataract surgery, using five response categories ranging from much lower to much higher (Longman 2012).
Decisional conflict | 2 weeks
  Decisional conflict will be measured using a scale named Decisional Conflict Scale. The scale is made of 16 items, using five response scores ranging from 0 to 4. The lower values represent a better outcome.
Decisional confidence | 2 weeks
  Decisional confidence will be assessed using a 11-item Decision Self Efficacy Scale.
Time perspective | 2 weeks
  This will be assessed using a 4-item short form of the Consideration of Future Consequences Scale, with five response categories ranging from strongly agree to strongly disagree.
Anticipated regret | 2 weeks
  Two items from a validated scale will measure anticipated regret about having cataract surgery (action regret) and about not having cataract (inaction regret).
Cataract worry and anxiety | 2 weeks
  A validated single item will measure participants' level of worry about progression of cataract , using four verbal response categories ranging from not worried at all to very worried. Anxiety will be measured with a six-item short form.
Booklet utilization and acceptability | 2 weeks
  We examined the utilization and acceptability of the decision aid using closed and open ended questions. Perceptions of the decision aid, in terms of its length, clarity, balance and usefulness in decision making were elicited using a modified scale (Mathieu 2010) (Smith 2009). We also asked participants to comment on their design preferences towards the booklets.
Undergoing cataract surgery | 1 year
  Self-reported undergoing cataract surgery will be assessed via telephone survey at 1 year.
Decision regret | 1 year
  The Decision Regret Scale will measure participants' level of regret regarding their initial decision whether to have cataract surgery or not.

CONTACTS AND LOCATIONS:
Overall Officials: Yingfeng Zheng, M.D. Ph.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen Univeristy
Locations (11):
- China (11):
  - Dashi Community Health Center, Guangzhou
  - Donghuan Community Health Center, Guangzhou
  - Huangcun Community Health Center, Guangzhou
  - Huaying Community Health Center, Guangzhou
  - Qiaonan Community Health Center, Guangzhou
  - Shawan Community Health Center, Guangzhou
  - Shibi Community Health Center, Guangzhou
  - Shiqiao Community Health Center, Guangzhou
  - Xiayuan Community Health Center, Guangzhou
  - Yuancun Community Health Center, Guangzhou
  - Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou

IPD SHARING:
Plan to Share IPD: No